CLINICAL TRIAL: NCT01129063
Title: An Open-label, Two-treatment Crossover Pharmacokinetic Study of Clopidogrel Hydrogen Sulfate in Healthy Male and Female Subjects
Brief Title: Pharmacokinetic Study of Single Doses of Clopidogrel, 75 mg and 300 mg, in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: International Clinical Development Study Director, sanofi-aventis
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PKM11086; 2008-008450-22 (EudraCT Number)
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequence clopidogrel 75 / 75 / 300 mg (Experimental): Period 1: clopidogrel 75 mg single dose
  Period 2: clopidogrel 75 mg single dose
  Period 3: clopidogrel 300 mg single dose
  Each intake is at around 8:00 AM under fasted conditions.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Pharmaceutical form : tablet
  Route of administration: oral
  Other Names: SR25990

SUMMARY:
The objectives of the study are to:

* Assess the within-subject variability of the pharmacokinetic profiles of the clopidogrel and its active metabolite after a replicated single administration of 75 mg of clopidogrel in healthy male and female subjects
* Assess the pharmacokinetic profiles of the clopidogrel and its active metabolite after single administration of 75 or 300 mg of clopidogrel

DETAILED DESCRIPTION:
The total study duration per subject is 4 - 6 weeks broken down as follows:

* Screening: 2 to 21 days before the first dosing
* Period 1, 2 and 3: 4 days including 1 treatment day each
* Washout between periods: at least 7 days between 2 administrations
* End of study: 7 to 10 days after the last dosing

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* as determined by medical history and complete physical examination including vital signs and clinical laboratory tests
* with a body weight between 50kg and 95 kg if male, between 40.0 kg and 85.0 kg if female and a Body Mass Index (BMI) between 18 and 28 kg/m2

Exclusion Criteria:

* Evidence of inherited disorder of coagulation/hemostasis functions
* Smoking more than 5 cigarettes or equivalent per day
* Abnormal hemostasis screen
* Any contraindication to clopidogrel
* Unability to abstain from intake of any drug affecting haemostasis throughout the whole study duration.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Clopidogrel pharmacokinetic parameters (Maximum plasma concentration (Cmax), Area under the plasma concentration curve (AUClast and AUC)) | Up to 48 hours postdose for each period
Clopidogrel active metabolite pharmacokinetic parameters (Cmax, AUClast and AUC) | Up to 48 hours postdose for each period

SECONDARY OUTCOMES:
Other clopidogrel pharmacokinetic parameters (first time to reach Cmax (tmax), terminal half-life (t1/2z)) | Up to 48 hours postdose for each period
Other clopidogrel active metabolite pharmacokinetic parameters (tmax, t1/2z) | Up to 48 hours postdose for each period

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development Study Director, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Paris, France